CLINICAL TRIAL: NCT04492904
Title: Singapore COVID-19 Chemosensory Tracking (SCCT) Study
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Vicki Tan, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2020/00810
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: Olfactory dysfunction; Gustatory dysfunction; Anosmia; Ageusia; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19; Anosmia; Ageusia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive (Case): Participants who were present for COVID-19 screening and their test results will later indicate positive of infection. Participants will complete a one-time assessment of the various online questionnaires (Singapore Smell and Test Questionnaire, Sino-nasal Outcome Test-22, and Global Consortium for Chemosensory Research Questionnaire - Optional) in the hospital/clinic. Taste and smell acuity, as well as experienced symptoms, changes in appetite and food-related quality of life will be assessed using the Home-use Tests and Follow-up questionnaire over a period of 28 days.
  Interventions: Other: Home-use Test and Follow-up Questionnaire
- COVID-19 Negative/Other respiratory diseases (Control): Participants who were present for COVID-19 screening and their test results will later indicate negative of infection. Participants will complete a one-time assessment of the various online questionnaires (Singapore Smell and Test Questionnaire, Sino-nasal Outcome Test-22, and Global Consortium for Chemosensory Research Questionnaire - Optional) in the hospital/clinic. Taste and smell acuity, as well as experienced symptoms, changes in appetite and food-related quality of life will be assessed using the Home-use Tests and Follow-up questionnaire over a period of 28 days
  Interventions: Other: Home-use Test and Follow-up Questionnaire

INTERVENTIONS:
Other: Home-use Test and Follow-up Questionnaire — Prospective tracking of changes in taste and smell acuity, and related changes in appetite, enjoyment of food and food-related quality of life will be assessed using the Home-use Tests and Follow-up questionnaire over a period of 28 days.

SUMMARY:
The study aims to longitudinally track the onset, severity and recovery of changes in chemosensory acuity (smell and/or taste loss) among those suspected of COVID-19 infection. Using standardised questionnaire and testing approaches, the investigators aim to objectively characterise and measure temporal changes in taste and smell to confirm the prevalence of these symptoms as an early marker of infection. Information on symptoms experience, changes in appetite and food-related quality of life will be also be assessed via questionnaire.

The results of the study will help individuals who experience a loss of smell and/or taste to self-isolate and/or self-refer to a medical professional, if an association between smell and/or taste and COVID-19 infection is found.

DETAILED DESCRIPTION:
The study will be a retrospective-prospective, longitudinal case-control observational study using a convenience sample drawn from patients presenting for COVID-19 screening, and will recruit both males and females above the age of 21 years who consent to provide anonymised data online on recent changes to their taste and smell. There will be no intervention (medication or foods) as part of this study. Potential participants will be screened to ensure they meet the study inclusion and exclusion criteria and all participants will sign an informed consent.

During their first recruitment session at the hospital/clinic, participants will be required to complete a series of questionnaires to record recent changes in taste and smell sensitivity. The series of questionnaires will include: Singapore Smell and Taste Questionnaire (SSTQ), Sino-nasal Outcome Test-22 (SNOT-22) and optionally, the Global Consortium of Chemosensory Research Questionnaire (GCCRQ). The purpose of administering the different questionnaires is to cover wide range of complementary questions that capture information related to changes in taste and smell function associated with COVID-19 infection. Thereafter participants will be briefed on how to complete the home-use standardized smell and taste test (Home-use Test). The Home-use Test (HUT) will be completed daily over a 28 day period at participants place of residence, to enable self-monitoring of changes to smell and taste abilities. During the HUT, participants will rate their sense of smell using the two standardised odour pens they are provided on the first day of their session at the hospital/ clinic. For each pen, participants will be asked to identify the odour and rate the perceived intensity. This will then be followed a taste test where participants will take a small quantity of a powder representing each of the four prototypical basic tastes sweet (sugar), salt (table salt), bitter (coffee powder or tea) and sour (lime powder), to the tip end of their tongue with a small spoon to taste. Participant are asked to self-report that they confirm that can identify the taste quality and to rate the perceived intensity on line scales provided in an online questionnaire. All measures are self-administered and completed independently by the participant, with responses captured using unique identifier code for each participant through an online software (CompuSense, Guelph, Ontario). During the 28-day home use test period, once a week participants will be asked to complete a 'Follow-up Questionnaire' which will assess how the symptoms experienced have impacted their enjoyment of food, appetite and food-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and above
* Residing in Singapore for the next 28 days.
* Possess a mobile device with 4G network and knows how to use mobile apps (i.e. QR scanner)

Exclusion Criteria:

* Unable to provide informed consent
* Allergic/ intolerant to test items (i.e. fragrances, sugar, salt, coffee or lime powder)
* Not agreeable with the study team accessing your medical records
* For women: Pregnant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients present for COVID 19 screening
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Taste and smell acuity | 28 days
  Taste and smell functions of all participants will be assessed as part of the Home-use Test using taste test items (i.e. sweet: sugar, salty: salt, sour: lime powder and bitter: coffee powder) and odour pens respectively. Participants will identify the taste/smell and rate the perceived intensity on a Visual Analogue Scale (VAS) from 'not strong at all' (0) to 'extremely strong taste/smell' (100). A higher score will indicate greater intensity of taste/smell perceived.

SECONDARY OUTCOMES:
Experienced symptoms, changes in appetite and food-related quality of life | 28 days
  Experienced symptoms, changes in appetite and food-related quality of life will be assessed as part of the Follow-up questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Forde, Phd, Principal Investigator — Singapore Institute of Food and Biotechnology Innovation
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Sheen F, Tan V, Haldar S, Sengupta S, Allen D, Somani J, Chen HY, Tambyah P, Forde CG. Evaluating the Onset, Severity, and Recovery of Changes to Smell and Taste Associated With COVID-19 Infection in a Singaporean Population (the COVOSMIA-19 Trial): Protocol for a Prospective Case-Control Study. JMIR Res Protoc. 2020 Dec 31;9(12):e24797. doi: 10.2196/24797. PMID 33351775